CLINICAL TRIAL: NCT00880789
Title: Adoptive Transfer of Cord Blood T Cells To Prevent and Treat CMV and Adenovirus Infections After Transplantation
Brief Title: Safety, Toxicity and MTD of One Intravenous IV Injection of Donor CTLs Specific for CMV and Adenovirus
Acronym: ACT-CAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Caridad Martinez, Prinicipal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23668-ACT CAT; NCT01017705 (obsolete NCT alias)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Cytomegalovirus Infection; Adenovirus Infection
Keywords: Cord Blood Transplant; cytomegalovirus; CMV; Adenovirus; ADV
MeSH Terms: conditions — Cytomegalovirus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Level One: 5x10^6/m2 (Experimental): CTL Dose Given from Day +30 post SCT (stem cell transplant). For the trial, two patients are allocated in each cohort and are followed for 30 days post IV injection of transduced T-cells for evaluation of DLTs. A maximum 18 patients will be accrued into each group. The final MTD will be the dose with probability closest to the target toxicity rate at these termination points. The trial continues until a minimum of 12 patients have been treated. The trial will stop when the maximum 18 patients have been treated, or when six patients have been treated at the current MTD. We therefore expect to enroll between 12-18 patients into this trial.
  Interventions: Biological: CMV/AdV specific T cells

INTERVENTIONS:
Biological: CMV/AdV specific T cells — CTL Dose Given from Day +30 post SCT (stem cell transplant). For the trial, two patients are allocated in each cohort and are followed for 30 days post IV injection of transduced T-cells for evaluation of DLTs. A maximum 18 patients will be accrued into each group. The final MTD will be the dose with probability closest to the target toxicity rate at these termination points. The trial continues until a minimum of 12 patients have been treated. The trial will stop when the maximum 18 patients have been treated, or when six patients have been treated at the current MTD. We therefore expect to enroll between 12-18 patients into this trial.

SUMMARY:
With this study, we want to see if we can use a kind of white blood cell called T cells to prevent or treat AdV and CMV infection. We will grow these T cells from the cord blood before the patients transplant. These cells have been trained to attack adenovirus/CMV-infected cells and are called Adenoviral/CMV-specific cytotoxic (killer) T-cells or "AdV/CMV-CTL." We would plan to give the patient one dose of AdV/CMV-CTL any time from 30 days after their transplant. We have used T cells made in this way from the blood of donors to prevent infections in patients who are getting a bone marrow or blood stem cell transplant but this will be the first time we make them from cord blood.

DETAILED DESCRIPTION:
We plan to grow T cells from the cord blood in the laboratory in a special way, to see if they can help prevent or treat infections in transplant patients with these viruses. This therapy with specially trained T cells (called CTLs) has had activity against these viruses when the cells are made from donor blood and given to patients receiving bone marrow or blood stem cell transplants. We want to find out if we can use CTLs that we will make from cord blood to prevent or treat viral infections when the patient's immunity is weak after receiving the cord blood transplant. These cells are called "CMV/AdV specific CTLs" because they can attack those two viruses.

The doctor will already have found a cord blood unit that is suitable for the patient's transplant. If the patient agrees to this study we will take 5-10 ml (1-2 teaspoons) from this cord blood unit before the transplant. We will only take as much cord blood as is available in a specially frozen small fraction of the cord blood unit.

We will use this cord blood to grow T cells in the lab. From this blood we will first grow special type of cells called dendritic cells and we will put a specially produced human virus (adenovirus) that carries the CMVpp65 gene into these dendritic cells. The dendritic cells will be irradiated so they cannot grow and then used to stimulate the T cells. This stimulation will train the T cells to kill cells with CMV and adenovirus on their surface.

We will then grow large numbers of these AdV/CMV-specific CTLs by more stimulation with EBV infected B cells (which we will make from the cord blood by infecting them with EBV in the laboratory). We will also put the special virus into these B cells so that they too have AdV/CMV. Again, these B cells will be treated with radiation so they cannot grow. Once we have made enough T cells we will test them to make sure they kill cells infected with Adenovirus and CMV. To make sure that these cells won't attack the patient's own healthy tissues, we test these cells against some of the blood cells that we will grow in the laboratory. These will be used to check to see if the AdV/CMV CTL can attack them. Alternatively, we may take blood from a first degree relative or take a small piece of skin from the patient to grow skin cells, which can also to be used to check if AdV/CMV CTL can attack them. The skin biopsy can be done at the same time as another procedure such as a bone marrow biopsy.

The cord donor's AdV/CMV CTL cells will be thawed and injected into the IV line over a period of up to 10 minutes.Patients may be premedicated with Benadryl and Tylenol. If the patient agrees and if he/she is well enough, one dose of CTL will be given on or after day 30 following transplant. If the patient does not have AdV/CMV infection we will not give antiviral medications to them during this study but we will monitor the patient closely to check for AdV/CMV infection. If the patient does have AdV/CMV infection before CTL infusion they may also be treated with antiviral medications during this study. We will monitor the patients closely for AdV/CMV infection by collecting blood and possibly urine and stool and testing them for AdV/CMV.

ELIGIBILITY:
INCLUSION CRITERIA:

Inclusion criteria at the time of Procurement:

* Patient with malignant or nonmalignant diseases who are candidates for transplant.
* Patients must have a single CB unit matched with the patient at 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens. The unit must be cryopreserved in two fractions, with a minimum of 2.5x10^7 total nucleated cells per kg pre-thaw in the fraction which will be used for the primary transplant. The remaining fraction will be used to generate the CTLs to give at day 30 or beyond as described below.

Inclusion criteria at the time of CTL infusion:

* Recipients of a single cord blood unit fractionated into 2 fractions (i.e. from a HLA matched or mismatched unrelated donor) transplant at risk for or with CMV/Adenoviral disease or reactivation.
* Lansky/Karnofsky scores 60 or greater
* Absolute neutrophil count (ANC) greater than 500/ul.
* No evidence of GVHD > Grade II at time of enrollment.
* Life expectancy > 30 days
* Absence of severe renal disease (Creatinine > x 3 normal for age)
* Absence of severe hepatic disease. Direct bilirubin must be less than 3 mg/dl and AST less than 5x upper limit of normal
* Patient must be at least 30 days post transplant to be eligible to receive CTL
* Written informed consent and/or signed assent line from patient, parent or guardian.
* Patient not on Fi02 of >60%

EXCLUSION CRITERIA:

Exclusion criteria at the time of Procurement:

* Pregnant or Lactating
* Patients with active central nervous system disease
* Patients with Karnofsky performance status <70%
* Patients with grade 3 or 4 or primary myelofibrosis
* Patients with suitable related donors

Exclusion criteria at the time of CTL infusion:

* Pregnant or lactating
* Unable to wean steroids to 0.5 mg/kg/day or less prednisone.
* Patients with other uncontrolled infections (except CMV and/or adenovirus and/or EBVemia in absence of PTLD). For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Patients with less than 50% donor chimerism in either peripheral blood or bone marrow or patients with relapse of original disease.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-05; Primary Completion 2013-08 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To determine safety, toxicity and MTD of one intravenous injection of donor-derived cytotoxic T lymphocytes (CTLs) specific for CMV and Adenovirus given to patients with or at risk for CMV and adenovirus disease after cord blood transplant | 1 year

SECONDARY OUTCOMES:
To evaluate the feasibility of generating a sufficient number of umbilical cord blood-derived cytotoxic T lymphocytes (CTLs) specific for CMV and Adenovirus | 1 year
To evaluate the impact of these CTLs on Adenovirus-specific T-lymphocyte immune reconstitution. | 1 year
To evaluate the recovery of virus-specific immunity after CTL infusion and its correlation with viral clearance and/or protection from viral infection/disease. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Caridad A. Martinez, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas